CLINICAL TRIAL: NCT04115397
Title: Towards Efficient Prediction and Prevention of Rheumatoid Arthritis
Brief Title: Bisphosphonates for the Treatment of Seropositive Musculoskeletal Complaints
Acronym: PREVENT RA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Anca Catrina, MD, PhD, Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2018/682-31
Record Dates: First submitted 2019-10-02; First posted 2019-10-04 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: Seropositive Muskuloskeletal Complaints
MeSH Terms: interventions — Zoledronic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bisphophonate (Experimental): Zolendronic acid, one infusion iv
  Interventions: Drug: Zoledronic Acid
- Placebo (Placebo Comparator): Placebo, one infusion iv
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Zoledronic Acid — Treating seropositive individuals with musculoskeletal symptoms with one infusion zolendronic acid as compared to placebo
  Arms: Bisphophonate
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Seropositive Rheumatoid arthritis (RA) is characterized by autoantibodies that develop prior to clinical onset, allowing identification of individuals at risk for disease development. In a unique program in Stockholm, seropositive individuals presenting with musculoskeletal complains are currently identified and followed-up in a dedicated outpatient clinical program. Despite significant disease burden and increased sick leave among these individuals, we lack today any therapeutic and preventive measures.

We aim to (1). establish a nation-wide health program, (2). develop an algorithm for disease risk estimation and (3). test a novel strategy to delay and/or prevent disease onset in seropositive at risk individuals with musculoskeletal complains. We will perform a multicentre randomised study to treat autoantibody-positive individuals at risk for developing RA presenting with pain (Population), by repurposing of bisphosphonates (Intervention) as compared to placebo (Control) to treat pain (primary Outcome) and delay/prevent RA development during 1-year follow-up (secondary Outcome)

DETAILED DESCRIPTION:
we have recently identified a novel disease-triggering pathogenic mechanism in autoantibody-positive individuals consisting in a bone-mediated induction of pain by autoantibodies. We hypothesize that specific targeting of this new mechanism, rather than using therapies developed for already established disease (where other mechanisms are active), will be able to treat pain with arthralgia and halt disease progression in seropositive at-risk individuals.

We will address this hypothesis by repurposing of bisphosphonates, currently used in clinical practice in both RA patients as well as in many individuals at risk for RA (mainly women in post-menopausal age). We will perform a multi centre, prospective, randomised, double-blind and placebo-controlled study with 2 parallel groups.

Patients will be randomised 1:1 to receive either one infusion aclasta (5 mg zolendronic acid, n=40) or placebo (n=40). The primary outcome is the VAS pain score and the study is powered to detect a 20% difference in the primary endpoint between the active and the control arm. The study is powered to detect a 20-percentage point difference in proportions between the control and the treated group. Subjects may withdraw from the trial at any time at their own or the investigators request for safety reasons.

ELIGIBILITY:
Inclusion Criteria:

Age older than 18 years Lack of arthritis as estimated by clinical and ultrasound examination of the joints ACPA positive Intermediate or high risk for RA (according to the algorithm described above) VAS score of at least 20 mm

Exclusion Criteria:

A previous diagnosis of arthritis Intolerance/contraindication to any of the study medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
VAS pain | 3 months
  PAin on a visual analogue scale

SECONDARY OUTCOMES:
HAQ | 3 months
  Health assessment questionnaire
MRI | 6 months
  MRI investigation of the symptomatic joints in the hands
Rheumatoid Arthritis (RA ) diagnosis | 1 year
  Getting a diagnosis of RA

IPD SHARING:
Plan to Share IPD: No